CLINICAL TRIAL: NCT06119269
Title: Ponatinib in cHronic myelOid LEukemia patieNts In Chronic phaSe: the PHOENICS Protocol
Brief Title: Ponatinib in Chronic Myeloid Leukemia Patients in Chronic Phase
Acronym: PHOENICS
Status: Recruiting | Type: Observational
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Antonello Di Paolo, M.D., Ph.D., Professor of Pharmacology, University of Pisa
Other Study IDs: 23707
Record Dates: First submitted 2023-10-18; First posted 2023-11-07 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Chronic Myeloid Leukemia, Chronic Phase
Keywords: Chronic myeloid leukemia, chronic phase; Ponatinib; Therapeutic drug monitoring; Efficacy; Tolerability
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase | interventions — Drug Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Therapeutic drug monitoring — At each follow up visit, plasma concentrations of ponatinib will be measured and compared with therapeutic range (according to a lower concentration equal to 21 nM)
Diagnostic Test: Molecular Response — BCR-ABl transcript levels will be assessed to evaluate molecular response to ponatinib

SUMMARY:
The goal of this retrospective observational study is to evaluate any possible association between plasma concentrations of ponatinib and its pharmacodynamics (efficacy/tolerability) in patients affected by chronic myeloid leukemia in chronic phase (CML-CP).

In particular, the aims of the study will be:

* primary aim: to investigate the relationships (if any) between plasma concentrations and activity/toxicity of ponatinib in a population of CML-CP patients enrolled in several Italian hematological centers;
* secondary aim: to set up an algorithm aimed at helping physicians to improve drug dosing based on several variables (i.e., plasma drug concentrations, tolerability, molecular response to therapy).

The study will enroll CML-CP patients who were exposed to ponatinib as second, third or fourth line of chemotherapy.

DETAILED DESCRIPTION:
The study protocol is a non-interventional, retrospective observational study which involves the collection of data from medical records relating to the plasma dosages of ponatinib performed as per clinical practice, all carried out at the pharmacokinetics laboratory of the Unit of Clinical Pharmacology and Pharmacogenetics of Azienda Ospedaliero Universitaria Pisana (AOUP). These data will be collected in CRF and will be correlated to efficacy data (extent of molecular response) and toxicity of ponatinib (haematological, extra-haematological adverse events, together with adverse event severity). Real-life experience (dosage adjustments made by clinicians based on plasma dosage) will be used to propose an algorithm that can help in choosing the correct dosage of ponatinib.

Classical statistical analyses (for descriptive and comparison aims) will be used according to their appropriateness. Moreover, factors affecting the pharmacokinetics (PK) of ponatinib will be investigated by nonlinear mixed effect modeling adopting the MONOLIX 2021R2 suite. Final model will be used as parte of the dosing algorithm.

Notably, all clinical and laboratory data will be anonymized to protect patients' privacy, and harvested in a database that will be used to perform pharmacometric and statistical analyses.

ELIGIBILITY:
Patients will be enrolled according the following inclusion criteria:

* Subjects ≥18 years old affected by CML
* Patients being treated with ponatinib at a dose of 45, 30 or 15 mg/day for more than 14 days
* Patients who have provided informed consent to the study

Exclusion criteria:

* Subjects <18 years old
* Patients who did not provide an informed consent to the study

The co-administration of drugs other than ponatinib will not be considered an exclusion criterium, but all of the drugs will be registered (together with daily doses and duration of treatment) as possible factors of ponatinib PK variability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with CML-CP who received ponatinib as 2nd-4th chemotherapy line will be enrolled according to inclusion/exclusion criteria listed.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-08-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Ponatinib plasma concentrations | 2 year
  Plasma concentrations of ponatinib included in the therapeutic range (i.e., >21 nM)

SECONDARY OUTCOMES:
Molecular response | Up to 2 year
  Plasma levels of BCR-ABl transcript
Occurrence of adverse events/adverse drug reactions | Up to 2 year
  Adverse events/Adverse drug reactions observed and registered during ponatinib administration

CONTACTS AND LOCATIONS:
Overall Officials: Sara Galimberti, PhD, Principal Investigator — University of Pisa - Dept. Clinical and Experimental Medicine
Locations (5):
- Italy (5):
  - University of Cagliari - Businco Hospital - Unit of Hematology and Bone Marrow Transplant, Cagliari
  - Policlinico Milano, Milan
  - University of Naples Federico II - Unit of Hematology, Napoli
  - Santa Chiara University Hospital, Pisa
  - Ospedale S. Eugenio ASL 2 Roma, Roma

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Galimberti S, Abruzzese E, Luci G, Barate C, Luciano L, Iurlo A, Caocci G, Morganti R, Stefanelli F, Di Paolo A. A New Algorithm Integrating Molecular Response, Toxicity, and Plasma Level Measures for Ponatinib Dose Choice in Patients Affected by Chronic Myeloid Leukemia. Pharmaceutics. 2024 Mar 11;16(3):383. doi: 10.3390/pharmaceutics16030383. PMID 38543276